CLINICAL TRIAL: NCT01583413
Title: CDC Prevention Epicenters Wake Up and Breathe Collaborative
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Pilgrim Health Care (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Washington University School of Medicine (Other); Rush University Medical Center (Other); University of Pennsylvania (Other); Duke University (Other); North Shore Medical Center (Other)
Responsible Party: Principal Investigator, Michael Klompas MD, MPH, FRCPC, Principal Investigator, Harvard Pilgrim Health Care
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH000410A-2; 3U54CK000172-01S1 (NIH)
Record Dates: First submitted 2012-04-20; First posted 2012-04-24 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Ventilator-associated Pneumonia
Keywords: Ventilator-associated pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Serum Bactericidal Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Opt Out Protocol (Experimental)
  Interventions: Procedure: Daily SAT & SBT

INTERVENTIONS:
Procedure: Daily SAT & SBT — Nurse and/or respiratory therapist led daily awakenings from sedation (spontaneous awakening trial, or SAT) and daily performance of a spontaneous breathing trial (SBT) among mechanically ventilated, critically ill patients in participating ICUs.

SUMMARY:
Ventilator-associated pneumonia (VAP) is a common complication of mechanical ventilation associated with significant morbidity, including prolongation of mechanical ventilation and increased ICU and hospital length-of-stay. Numerous strategies have been proposed to decrease the occurrence of VAP among ventilated patients. Most notably, optimizing the use of daily sedative interruptions and daily spontaneous breathing trials can improve sedative management, decrease ventilator time, improve outcomes for mechanically ventilated patients,and possibly decrease VAP.Combining daily sedative interruption with daily spontaneous breathing trials confers additive improvement in ventilator days, intensive care days, and possibly mortality compared to daily spontaneous breathing trials alone.

The primary aim of this study is to determine the impact of an opt-out protocol for paired daily sedative interruptions and spontaneous breathing trials on VAP rates using a new streamlined VAP definition. The investigators will evaluate the responsiveness of CDC's proposed new surveillance definitions for ventilator-associated events to this quality improvement initiative. The study will be nested within the Epicenters Streamlined versus Conventional VAP Surveillance Study. Nine of the 18 hospitals in the larger study will be participating in this intervention arm.

ELIGIBILITY:
Inclusion Criteria:

* all patients in participating units on mechanical ventilation for at least one calendar day beting treated with continuous sedatives or standing orders for sedatives. Patients receiving mechanical ventilation through either an endotracheal or tracheostomy tube will be eligible.

Exclusion Criteria:

* moribund status or plans for withdrawal of life support

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3342 (Actual)
Dates: Start 2012-05; Primary Completion 2013-06 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change in VAC rate. | 12 months
  A new definition for VAP is the primary focus of this study. This new definition (referred to as "streamlined VAP" or "sVAP") is under consideration by the CDC as a potential replacement for the current NHSN VAP definition and, as such, will be closely evaluated to determine if it can reflect meaningful changes in patient care. Thus, we will assess the change in monthly sVAP rates from study start to study end using an interrupted time series analysis.
  Note that CDC released new surveillance definitions for ventilator-associated events in late 2012. Given that CDC definitions are the defacto surveillance standard, we switched the primary study outcome from sVAP to ventilator-associated conditions ("VAC"). All data elements required to assess for VAC were included in this study from the outset hence we did not have to collect any additional historical data in order to apply CDC's VAC definition.

SECONDARY OUTCOMES:
ICU-specific outcomes | 12-months
  * NHSN VAP rate
  * Mechanical ventilation days per patient
  * Ventilator-free days assessed over 28 days post-intubation
  * ICU length of stay per patient
  * Average antibiotic days
  * Rates of extubation and reintubation within 48 hours
Hospital-specific outcomes | 12-months
  * Hospital length of stay
  * Hospital mortality
Patient-specific outcomes | 12-months
  * Mean ventilator days
  * Mean ICU days
  * Mean hospital days
  The above results will also be assessed separately for patients who received opt-out protocol care versus those who did not.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Klompas, MD, MPH, Principal Investigator — Harvard Pilgrim Health Care
Locations (5):
- United States (5):
  - Chicago Prevention Epicenter, Chicago, Illinois
  - North Shore Medical Center, Salem, Massachusetts
  - Washington University Prevention Epicenter, St Louis, Missouri
  - Duke University Prevention Epicenter, Durham, North Carolina
  - University of Pennsylvania Prevention Epicenter, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Klompas M, Anderson D, Trick W, Babcock H, Kerlin MP, Li L, Sinkowitz-Cochran R, Ely EW, Jernigan J, Magill S, Lyles R, O'Neil C, Kitch BT, Arrington E, Balas MC, Kleinman K, Bruce C, Lankiewicz J, Murphy MV, E Cox C, Lautenbach E, Sexton D, Fraser V, Weinstein RA, Platt R; CDC Prevention Epicenters. The preventability of ventilator-associated events. The CDC Prevention Epicenters Wake Up and Breathe Collaborative. Am J Respir Crit Care Med. 2015 Feb 1;191(3):292-301. doi: 10.1164/rccm.201407-1394OC. PMID 25369558